CLINICAL TRIAL: NCT03577028
Title: A Phase 1/2a Open-label, Multicenter, Dose Escalation and Dose Expansion Study of the Safety, Tolerability, and Pharmacokinetics of HPN424 in Patients With Advanced Prostate Cancer Refractory to Androgen Therapy
Brief Title: Study of HPN424 in Patients With Advanced Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Decision not to continue to the expansion portion of the study
Sponsor: Harpoon Therapeutics, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HPN424-1001
Record Dates: First submitted 2018-06-22; First posted 2018-07-05 (Actual); Results first posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Advanced Prostate Cancer
Keywords: Prostate Cancer; Metastatic Castration Resistant Prostate Cancer; Harpoon; TriTAC
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Fixed IV (Experimental): HPN424 administered once weekly via IV infusion in doses ranging from 1.3 to 150 ng/kg
  Interventions: Biological: HPN424 Fixed IV 1.3 to 150 ng/kg
- 1 Prime Step IV 36 ng/kg Target (Experimental): Step-dosing IV cohort who received a single Prime Dose followed by the Target Dose (12/36 ng/kg)
  Interventions: Biological: HPN424 Prime Step IV 36 ng/kg Target
- 1 Prime Step IV 225-300 ng/kg Target (Experimental): Step-dosing IV cohorts who received a single Prime Dose followed by the Target Dose (100/300 ng/kg and 75/225 ng/kg]
  Interventions: Biological: HPN424 1 Prime Step IV 225-300 ng/kg Target
- 2 Prime Step IV 300 ng/kg Target (Experimental): Step-dosing IV cohorts who received 2 Prime Doses followed by the Target Dose (50/150/300 ng/kg with prior chemotherapy and 50/150/300 ng/kg no prior chemotherapy)
  Interventions: Biological: HPN424 2 Prime Step IV 300 ng/kg Target
- 2 Prime Step IV 450 ng/kg Target (Experimental): Step-dosing IV cohorts who received 2 Prime Doses followed by the Target Dose (100/300/450 ng/kg and 50/150/450 ng/kg)
  Interventions: Biological: HPN424 2 Prime Step IV 450 ng/kg Target
- Fixed SC (Experimental): Fixed subcutaneous dose (120 ng/kg)
  Interventions: Biological: HPN424 Fixed SC

INTERVENTIONS:
Biological: HPN424 Fixed IV 1.3 to 150 ng/kg — Fixed dose IV cohorts at doses from 1.3 to 150 ng/kg
  Arms: Fixed IV
Biological: HPN424 Prime Step IV 36 ng/kg Target — Step-dosing IV cohort at a single Prime Dose followed by the Target Dose (12/36 ng/kg)
  Arms: 1 Prime Step IV 36 ng/kg Target
Biological: HPN424 1 Prime Step IV 225-300 ng/kg Target — Step-dosing IV cohorts who received a single Prime Dose followed by the Target Dose (100/300 ng/kg and 75/225 ng/kg)
  Arms: 1 Prime Step IV 225-300 ng/kg Target
Biological: HPN424 2 Prime Step IV 300 ng/kg Target — Step-dosing IV cohorts who received 2 Prime Doses followed by the Target Dose (50/150/300 ng/kg with prior chemotherapy and 50/150/300 ng/kg no prior chemotherapy)
  Arms: 2 Prime Step IV 300 ng/kg Target
Biological: HPN424 2 Prime Step IV 450 ng/kg Target — Step-dosing IV cohorts who received 2 Prime Doses followed by the Target Dose (100/300/450 ng/kg and 50/150/450 ng/kg)
  Arms: 2 Prime Step IV 450 ng/kg Target
Biological: HPN424 Fixed SC — Fixed subcutaneous dose 120 ng/kg
  Arms: Fixed SC

SUMMARY:
An open-label, Phase 1/2a, study of HPN424 as monotherapy to assess the safety, tolerability and PK in patients with advanced prostate cancer refractory to androgen therapy

ELIGIBILITY:
Inclusion Criteria:

1. Male patients ≥18 years of age at the time of signing informed consent
2. Histologically or cytologically confirmed adenocarcinoma of the prostate
3. Progressive metastatic castrate-resistant prostate cancer (mCRPC):

   1. Serum testosterone levels less than 50 ng/dL (or ≤0.50 ng/mL or 1.73 nmol/L) within 28 days prior to start of study drug
   2. Radiographic evidence of metastatic disease
   3. Disease progression on the prior systemic regimen, per Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria:

   i. A sequence of at least 2 rising PSA values measured at a minimum of 1 week apart with a 2 ng/mL minimum starting value, or ii. Appearance of two or more new lesions on bone scans, or iii. Progressive visceral disease, or iv. Progressive nodal disease; previously normal (<1.0 cm) lymph nodes must have grown by ≥5 mm in the short axis from baseline or nadir and be ≥1.0 cm in the short axis to be considered to have progressed
4. Must have received at least 2 prior systemic therapies approved for mCRPC
5. Ongoing androgen depletion therapy with a gonadotropin releasing hormone analog or inhibitor, or orchiectomy (surgical or medical castration)
6. For patients previously treated with first generation anti-androgens, discontinuation must have occurred ≥4 weeks (for flutamide or nilutamide) or ≥6 weeks (for bicalutamide) prior to start of study drug, with no evidence of an anti-androgen withdrawal response (i.e., no decline in serum PSA)
7. For patients previously treated with a second-generation anti-androgen (e.g., enzalutamide or equivalent) or with abiraterone acetate, discontinuation must have occurred 2 weeks or 5 half-lives prior to start of study drug
8. For patients previously treated with systemic chemotherapy, targeted therapy, immunotherapy, or treatment with an investigational anticancer agent, discontinuation must have occurred ≥2 weeks, or at least 4 half-lives (up to 4 weeks), whichever is longer, prior to start of study drug
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
10. Adequate bone marrow function, including:

    1. Absolute neutrophil count (ANC) ≥1500/mm3 or ≥1.5 x 109/L
    2. Platelets ≥100,000/mm3 or ≥100 x 109/L
    3. Hemoglobin ≥9 g/dL (no transfusions allowed within 1 week prior to screening)
11. Adequate renal function, including:

    a. Estimated creatinine clearance ≥50 mL/min as calculated using the method standard for the institution
12. Adequate liver function, including:

    1. Total serum bilirubin ≤1.5 x upper limit of normal (ULN) unless the patient has documented Gilbert syndrome in which case the maximum total serum bilirubin should be 5 mg/dL
    2. Aspartate and Alanine transaminase (AST and ALT) ≤2.5 x ULN
13. Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade ≤1 except for adverse events (AEs) not constituting a safety risk per the Investigator
14. If of reproductive potential, willing to use 1 effective method of contraception (as defined in this protocol) during the treatment period, if partner is a female of childbearing potential
15. Willing to complete all scheduled visits and assessments at the institution administering therapy
16. Able to read, understand and provide written informed consent

Exclusion Criteria:

1. Previously treated or current brain metastases
2. Untreated spinal cord compression. Participants must be neurologically stable off steroids for at least 4 weeks prior to first dose of study drug
3. Ongoing treatment with anti-tumor necrosis factor (TNF) alpha therapies, systemic corticosteroids (prednisone dose >10 mg per day or equivalent), or other immune suppressive drugs
4. History of or known or suspected autoimmune disease (exception(s): patients with vitiligo, resolved childhood atopic dermatitis, hypothyroidism, or hyperthyroidism that is clinically euthyroid at Screening are allowed)
5. History of clinically significant cardiovascular disease such as symptomatic congestive heart failure (CHF), uncontrolled hypertension defined as sustained BP >150 mmHg systolic, or >100 mmHg diastolic despite optimal antihypertensive treatment (BP must be controlled at screening), unstable angina pectoris, clinically significant cardiac arrhythmias, history of stroke (including TIA, or other ischemic event) within 6 months before first dose of study drug, myocardial infarction within 6 months before first dose of study drug, history of thromboembolic event within 3 months before first dose of study drug
6. Known active or chronic hepatitis B or hepatitis C as demonstrated by hepatitis B surface antigen (HBsAg) positivity and/or anti-hepatitis C virus (HCV) positivity, respectively, or known history of human immunodeficiency virus (HIV) seropositive status
7. Clinically active liver disease, including liver cirrhosis of Child-Pugh class B or C
8. Second primary malignancy that has not been in remission for greater than 3 years. Exceptions that do not require a 3-year remission: non-melanoma skin cancer, resected melanoma in situ, or non-muscle invasive urothelial carcinoma
9. In the judgment of the Investigator, patient has a clinically significant concurrent illness or psychological, familial, sociological, geographical, or other concomitant condition that would not permit adequate follow-up and compliance with the study protocol
10. Any serious underlying medical or psychiatric condition (e.g., alcohol or drug abuse), dementia or altered mental status or any issue that would impair the ability of the patient to understand informed consent or that in the opinion of the Investigator would contraindicate the patient's participation in the study or confound the results of the study
11. Known hypersensitivity, allergies, or intolerance to immunoglobulins, or to any excipient contained in HPN424 (see Investigator's Brochure)
12. Is a participant or plans to participate in another interventional clinical study, while taking part in this protocol. Participation in an observational study is acceptable

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (14):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Hospital, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - New York Presbyterian Hospital-Columbia University Medical Center., New York, New York
  - Oregon Health & Science University Knight Cancer Institute, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- The Royal Marsden Hospital, Sutton, Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Fixed IV: Fixed dose IV cohorts (1.3 to 150 ng/kg). The study was terminated early, therefore the primary goal of the final data analysis was to look at dosing schedule rather than individual dose levels. The results displayed are shown broken out by dosing schedules and no analysis of specific dose levels was performed. This analysis is as outlined in the final Statistical Analysis Plan.
- 1 Prime Step IV 36 ng/kg Target: Step-dosing IV cohort who received a single Prime Dose followed by the Target Dose (12/36 ng/kg). The study was terminated early, therefore the primary goal of the final data analysis was to look at dosing schedule rather than individual dose levels. The results displayed are shown broken out by dosing schedules and no analysis of specific dose levels was performed. This analysis is as outlined in the final Statistical Analysis Plan.
- 1 Prime Step IV 225-300 ng/kg Target: Step-dosing IV cohorts who received a single Prime Dose followed by the Target Dose (100/300 ng/kg and 75/225 ng/kg). The study was terminated early, therefore the primary goal of the final data analysis was to look at dosing schedule rather than individual dose levels. The results displayed are shown broken out by dosing schedules and no analysis of specific dose levels was performed. This analysis is as outlined in the final Statistical Analysis Plan.
- 2 Prime Step IV 300 ng/kg Target: Step-dosing IV cohorts who received 2 Prime Doses followed by the Target Dose (50/150/300 ng/kg with prior chemotherapy and 50/150/300 ng/kg no prior chemotherapy). The study was terminated early, therefore the primary goal of the final data analysis was to look at dosing schedule rather than individual dose levels. The results displayed are shown broken out by dosing schedules and no analysis of specific dose levels was performed. This analysis is as outlined in the final Statistical Analysis Plan.
- 2 Prime Step IV 450 ng/kg Target: Step-dosing IV cohorts who received 2 Prime Doses followed by the Target Dose (100/300/450 ng/kg and 50/150/450 ng/kg). The study was terminated early, therefore the primary goal of the final data analysis was to look at dosing schedule rather than individual dose levels. The results displayed are shown broken out by dosing schedules and no analysis of specific dose levels was performed. This analysis is as outlined in the final Statistical Analysis Plan.
- Fixed SC: Fixed subcutaneous dose 120 ng/kg. The study was terminated early, therefore the primary goal of the final data analysis was to look at dosing schedule rather than individual dose levels. The results displayed are shown broken out by dosing schedules and no analysis of specific dose levels was performed. This analysis is as outlined in the final Statistical Analysis Plan.
Period: Overall Study
Arm/Group | Fixed IV | 1 Prime Step IV 36 ng/kg Target | 1 Prime Step IV 225-300 ng/kg Target | 2 Prime Step IV 300 ng/kg Target | 2 Prime Step IV 450 ng/kg Target | Fixed SC
Started | 64 | 6 | 12 | 10 | 9 | 3
Completed | 64 | 6 | 12 | 10 | 9 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population. The study was terminated early, therefore the primary goal of the final data analysis was to look at dosing schedule rather than individual dose levels. The results displayed are shown broken out by dosing schedules and no analysis of specific dose levels was performed. This analysis is as outlined in the final Statistical Analysis Plan.
Groups:
- Fixed IV: Fixed dose IV cohorts (1.3 to 150 ng/kg)
- 1 Prime Step IV 225-300 ng/kg Target: Step-dosing IV cohorts who received a single Prime Dose followed by the Target Dose (100/300 ng/kg and 75/225 ng/kg)
- Fixed SC: Fixed subcutaneous dose 120 ng/kg
- Total: Total of all reporting groups
Arm/Group | Fixed IV | 1 Prime Step IV 36 ng/kg Target | 1 Prime Step IV 225-300 ng/kg Target | 2 Prime Step IV 300 ng/kg Target | 2 Prime Step IV 450 ng/kg Target | Fixed SC | Total
Number analyzed (Participants) | 64 | 6 | 12 | 10 | 9 | 3 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 0 | 6 | 3 | 2 | 0 | 25
  >=65 years | 50 | 6 | 6 | 7 | 7 | 3 | 79
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 64 | 6 | 12 | 10 | 9 | 3 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 0 | 1 | 0 | 4
  Not Hispanic or Latino | 55 | 6 | 10 | 10 | 7 | 3 | 91
  Unknown or Not Reported | 6 | 0 | 2 | 0 | 1 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Black or African American | 6 | 2 | 1 | 0 | 0 | 0 | 9
  White | 49 | 4 | 9 | 10 | 9 | 3 | 84
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 0 | 2 | 0 | 0 | 0 | 7
Region of Enrollment [Number; unit: participants]
  United States | 56 | 6 | 11 | 9 | 6 | 3 | 91
  United Kingdom | 8 | 0 | 1 | 1 | 3 | 0 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number and Severity of Dose Limiting Toxicities (DLTs) Following Treatment With Escalating Doses of HPN424
Description: Assess safety and tolerability at increasing dose levels of HPN424 in successive cohorts of patients with metastatic castrate resistant prostate cancer (mCRPC) to estimate the maximum tolerated dose (MTD). The study was terminated early, therefore the primary goal of the final data analysis was to look at dosing schedule rather than individual dose levels. The results displayed are shown broken out by dosing schedules and no analysis of specific dose levels was performed. This analysis is as outlined in the final Statistical Analysis Plan.
Time Frame: 21 days
Population: Safety population receiving at least one dose. The study was terminated early, and therefore the primary goal of the final data analysis was to look at dosing schedule rather than individual dose levels. The results displayed are shown broken out by dosing schedules and no analysis of specific dose levels was performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed IV | 1 Prime Step IV 36 ng/kg Target | 1 Prime Step IV 225-300 ng/kg Target | 2 Prime Step IV 300 ng/kg Target | 2 Prime Step IV 450 ng/kg Target | Fixed SC
Number analyzed (Participants) | 64 | 6 | 12 | 10 | 9 | 3
Participants | 6 | 0 | 4 | 2 | 3 | 1

ADVERSE EVENTS:
Time Frame: From 28 days after they received their last dose of study drug to study completion, a median of approximately 313 days. Participants continued to receive doses until they progressed or stopped treatment for other reasons.
Description: All events that occur or worsen in severity or frequency during or after the first HPN424 study drug administration through 28 days after the last dose of study drug. The primary goal of the final data analysis was to look at dosing schedule rather than individual dose levels. The results displayed are shown broken out by dosing schedules and no analysis of specific dose levels was performed. This analysis is as outlined in the final Statistical Analysis Plan.
Arm/Group | Fixed IV | 1 Prime Step IV 36 ng/kg Target | 1 Prime Step IV 225-300 ng/kg Target | 2 Prime Step IV 300 ng/kg Target | 2 Prime Step IV 450 ng/kg Target | Fixed SC
All-Cause Mortality (participants affected / at risk) | 37/64 | 3/6 | 9/12 | 5/10 | 3/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 41/64 | 3/6 | 7/12 | 8/10 | 5/9 | 1/3
Other Adverse Events (participants affected / at risk) | 64/64 | 6/6 | 12/12 | 10/10 | 9/9 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fixed IV (N=64) | 1 Prime Step IV 36 ng/kg Target (N=6) | 1 Prime Step IV 225-300 ng/kg Target (N=12) | 2 Prime Step IV 300 ng/kg Target (N=10) | 2 Prime Step IV 450 ng/kg Target (N=9) | Fixed SC (N=3)
Cytokine release syndrome (Immune system disorders) | 17 | 0 | 3 | 6 | 0 | 0
Type IV hypersensitivity reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 0 | 1 | 2 | 3 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0 | 1 | 1 | 3 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram ST-T segment abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 2 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fixed IV (N=64) | 1 Prime Step IV 36 ng/kg Target (N=6) | 1 Prime Step IV 225-300 ng/kg Target (N=12) | 2 Prime Step IV 300 ng/kg Target (N=10) | 2 Prime Step IV 450 ng/kg Target (N=9) | Fixed SC (N=3)
Fatigue (General disorders) | 33 | 4 | 8 | 6 | 6 | 2
Pyrexia (General disorders) | 18 | 1 | 0 | 5 | 1 | 0
Chills (General disorders) | 14 | 1 | 0 | 2 | 4 | 1
Oedema peripheral (General disorders) | 3 | 1 | 0 | 2 | 2 | 0
Asthenia (General disorders) | 7 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 2 | 1 | 2 | 0 | 0 | 0
Injection site reaction (General disorders) | 2 | 0 | 0 | 0 | 0 | 2
Pain (General disorders) | 2 | 0 | 0 | 1 | 1 | 0
Chest discomfort (General disorders) | 2 | 0 | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Catheter site extravasation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hernia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vascular device occlusion (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 22 | 0 | 6 | 8 | 9 | 1
Alanine aminotransferase increased (Investigations) | 21 | 0 | 7 | 8 | 8 | 1
Blood alkaline phosphatase increased (Investigations) | 5 | 0 | 2 | 2 | 5 | 2
Blood bilirubin increased (Investigations) | 8 | 0 | 3 | 1 | 3 | 0
Lymphocyte count decreased (Investigations) | 4 | 0 | 3 | 3 | 3 | 1
Blood creatinine increased (Investigations) | 8 | 1 | 1 | 1 | 1 | 0
Weight decreased (Investigations) | 5 | 0 | 3 | 3 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 3 | 0 | 3 | 2 | 1 | 1
Platelet count decreased (Investigations) | 2 | 0 | 3 | 1 | 4 | 0
White blood cell count decreased (Investigations) | 3 | 0 | 3 | 1 | 3 | 0
Blood calcium decreased (Investigations) | 2 | 0 | 2 | 1 | 2 | 0
Blood albumin decreased (Investigations) | 2 | 0 | 2 | 1 | 1 | 0
Blood sodium decreased (Investigations) | 2 | 0 | 2 | 1 | 1 | 0
C-reactive protein increased (Investigations) | 2 | 0 | 1 | 2 | 1 | 0
Neutrophil count decreased (Investigations) | 3 | 0 | 2 | 1 | 0 | 0
Blood glucose increased (Investigations) | 2 | 0 | 2 | 0 | 1 | 0
Amylase increased (Investigations) | 2 | 0 | 1 | 0 | 1 | 0
Blood phosphorus decreased (Investigations) | 2 | 0 | 0 | 1 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 2 | 0 | 1 | 0
Lipase increased (Investigations) | 2 | 0 | 0 | 1 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 2 | 1 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 1 | 1
Haematocrit decreased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0
Liver function test increased (Investigations) | 2 | 0 | 0 | 1 | 0 | 0
Mean cell haemoglobin concentration decreased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0
Red cell distribution width increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0
Amylase decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Platelet count increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Blood albumin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood chloride increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Carbon dioxide decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram ST-T segment abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Mean cell haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 23 | 2 | 5 | 3 | 4 | 1
Vomiting (Gastrointestinal disorders) | 14 | 3 | 6 | 3 | 3 | 0
Constipation (Gastrointestinal disorders) | 18 | 0 | 3 | 1 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 1 | 3 | 6 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 7 | 0 | 3 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 0 | 2 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0
Eructation (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lip blister (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 42 | 3 | 10 | 8 | 9 | 3
Type IV hypersensitivity reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 1 | 6 | 4 | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 0 | 3 | 3 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 0 | 1 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 0 | 0 | 1 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 7 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 0 | 3 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 15 | 1 | 4 | 3 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 0 | 1 | 3 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 1 | 0 | 0 | 3 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 1 | 1 | 1 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 0 | 0 | 1 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 2 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 23 | 2 | 3 | 5 | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 0 | 0 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 0 | 2 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Cytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 10 | 0 | 4 | 3 | 1 | 0
Dizziness (Nervous system disorders) | 10 | 0 | 1 | 1 | 2 | 0
Dysgeusia (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 4 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 2 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 1 | 2 | 1 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2 | 1 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 15 | 2 | 3 | 3 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 1 | 1
Hyphaema (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 0 | 2 | 2 | 0 | 0
COVID-19 (Infections and infestations) | 3 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Mastoiditis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Phlebitis infective (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Stoma site cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 9 | 1 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 5 | 0 | 0 | 3 | 2 | 1
Flushing (Vascular disorders) | 3 | 1 | 0 | 1 | 1 | 0
Hot flush (Vascular disorders) | 4 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 1 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 11 | 0 | 1 | 2 | 1 | 0
Confusional state (Psychiatric disorders) | 6 | 0 | 3 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 5 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 7 | 1 | 0 | 2 | 3 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 0 | 1 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 3 | 0 | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 1 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract discomfort (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 3 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Photopsia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Strabismus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Penile pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT03577028/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT03577028/SAP_001.pdf